CLINICAL TRIAL: NCT01580202
Title: A Randomized, Open Labeled, Multicenter Study Comparing Entecavir Versus Lamivudine as Antiviral Prophylaxis for Patients With Hepatitis B Infection Undergoing Cytotoxic Chemotherapy for Malignant Tumors
Brief Title: Comparison of Prophylactic Antiviral Efficacy in Patients Undergoing Chemotherapy: Entecavir Versus Lamivudine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sook-Hyang Jeong, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-246
Record Dates: First submitted 2012-04-04; First posted 2012-04-18 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Malignancy; Hepatitis B
Keywords: malignancy; hepatitis B; lamivudine; entecavir; prophylaxis
MeSH Terms: conditions — Neoplasms; Hepatitis B | interventions — entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamivudine (Active Comparator): LAM (100 mg/day) will be started within 1 week prior to initiation of the 1st cycle of chemotherapy, and continued until 24 weeks after completion of the last chemotherapy.
  Interventions: Drug: Lamivudine
- Entecavir (Experimental): ETV (0.5 mg/day) will be started within 1 week prior to initiation of the 1st cycle of chemotherapy, and continued until 24 weeks after completion of the last chemotherapy.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Entecavir 0.5mg daily per os
  Arms: Entecavir
Drug: Lamivudine — lamivudine 100mg daily per os
  Arms: Lamivudine

SUMMARY:
Patients with chronic hepatitis B who are undergoing anticancer chemotherapy are at risk of HBV reactivation and hepatitis flare. Lamivudine (LAM) prophylaxis has been recommended in such circumstance according to the practice guidelines despite of limited evidence. However, failure of LAM prophylaxis including virologic breakthrough and withdrawal hepatitis occurs occasionally, which may lead to liver-related morbidity and mortality as well as premature interruption or a delay of chemotherapy. Given relatively frequent drug resistance of LAM, studies on the proper prophylactic antiviral regimen is warranted. The present multicenter, prospective, randomized study aims to compare the effect of entecavir (ETV) versus LAM for the prevention of HBV reactivation in HBsAg-positive patients with hematologic and oncologic malignancy undergoing cytotoxic chemotherapy.

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) carriers who are undergoing anticancer chemotherapy are at risk of HBV reactivation and hepatitis flare, and lamivudine (LAM) prophylaxis is recommended according to the practice guidelines despite of limited evidence. However, failure of LAM prophylaxis defined as virologic breakthrough during LAM therapy and withdrawal hepatitis after discontinuation of LAM therapy occurs occasionally, which may lead to liver-related morbidity and mortality as well as premature interruption or a delay of chemotherapy. Considering that LAM therapy showed relatively higher rates of drug resistance and of withdrawal hepatitis, studies on the better choice of prophylactic antiviral regimen is warranted.

The purpose of our study is to conduct a multicenter, prospective, randomized study comparing the effect of entecavir (ETV) versus LAM for the prevention of HBV reactivation in HBsAg-positive patients with hematologic and oncologic malignancy undergoing cytotoxic chemotherapy.

A total one hundred eighty HBV carriers with malignancy undergoing chemotherapy will be randomly assigned to each prophylactic therapy arm of ETV and LAM group. The primary endpoint of the study is the HBV reactivation rate during antiviral therapy and 6 months after discontinuation of prophylactic antiviral therapy.

If the prophylactic efficacy of ETV is superior to that of LAM, ETV will be the preferred prophylactic therapy for HBsAg-positive cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* positive for HBsAg for at least 6 months
* inactive or active carrier of HBV with ALT level <2xULN, chronic hepatitis and compensated cirrhosis (Child-Pugh class A)
* malignant tumors: non-Hodgkin's lymphoma undergoing systemic chemotherapy; solid tumors undergoing chemotherapy (including adjuvant/neoadjuvant chemotherapy or concurrent chemoradiation therapy)

Exclusion Criteria:

* positive for anti-HCV or anti-HIV antibodies
* decompensated cirrhosis or hepatocellular carcinoma
* expected survival of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The cumulative probability of HBV reactivation | From the time of randomization until 24week after discontinuation of antiviral prophylaxis
  10-fold or more elevation in serum HBV DNA titers above nadir

SECONDARY OUTCOMES:
Incidence of HBV-related hepatitis flare | From the time of randomization until 24week after discontinuation of antiviral prophylaxis
  greater than 3-fold increase of ULN (upper limit of a normal reference value) of a serum ALT level that exceeded 100 IU/L during antiviral prophylaxis and 24 week after discontinuation of antiviral prophylaxis
Cumulative probability of emergence of genotypic resistance | From the time of randomization until 24week after discontinuation of antiviral prophylaxis
  detection of mutations that have been shown in in vitro studies to confer resistance to either ETV or LAM
Incidence of hepatic decompensation and liver-related mortality | From the time of randomization until 24week after discontinuation of antiviral prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Sook-Hyang Jeong, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (5):
- South Korea (5):
  - National Cancer Center, Korea, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si
  - Seoul National University Hospital, Seoul
  - Seoul National University Boramae Hospital, Seoul